CLINICAL TRIAL: NCT01948388
Title: Study of The Effect of Corticotrophin in Combination With Methotrexate in Newly Diagnosed Rheumatoid Arthritis Patients From a Clinical and Structural Perspective As Measured by a Clinical Disease Activity Index Score and Bone Edema, Synovitis and Erosions on Magnetic Resonance Imaging
Brief Title: The Effect of Corticotrophin (ACTH) in Combination With Methotrexate in Newly Diagnosed Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gaylis, Norman B., M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RA2013-01
Record Dates: First submitted 2013-09-09; First posted 2013-09-23 (Estimated); Results first posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- corticotrophin 80 units (Active Comparator): Ten (10) patients will receive 80 units of corticotrophin Subcutaneous (SC) weekly
  Interventions: Drug: corticotrophin 80 units
- corticotrophin 80 units twice a week (Active Comparator): Ten (10) patients will receive 80 units of corticotrophin Subcutaneous (SC) twice a week
  Interventions: Drug: corticotrophin 80 units

INTERVENTIONS:
Drug: corticotrophin 80 units — Comparison of different dosages of the drug. Ten patients will receive 80 units of corticotrophin weekly. Ten patients will receive 80 units bi-weekly of corticotrophin
  Other Names: Acthar, Corticotrophin, ACTH

SUMMARY:
The purpose of the study is to evaluate the effect of the utilization of two doses of corticotrophin ( ACTH) as a treatment in patients with early onset rheumatoid arthritis as an alternative to conventional steroid therapy by evaluating the change from baseline in the clinical findings as well as the structural findings on Magnetic Resonance Imaging (MRI). Corticotrophin (ACTH) may prevent the well documented structural progression damage in RA patients using disease-modifying antirheumatic drug (DMARD) therapy alone.

DETAILED DESCRIPTION:
This is a Phase II 24-week open-label study to evaluate the efficacy and safety of H.P. Acthar Gel Respository Injection, Corticotrophin( ACTH) administered to newly diagnosed patients with rheumatoid arthritis in conjunction with methotrexate, folllowed by a 24 week follow-up period. There will be a total of twenty (20) patients and two (2) treatment groups with 10 patients in each treatment group

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 18 years old at the screening visit.
2. Patient must be able to understand the information provided to them and to give written Informed Consent.
3. Female patients must be either postmenopausal for at least 1 year, surgically incapable of childbearing, or effectively practicing an acceptable method of contraception (oral/parenteral/implantable hormonal contraceptives, Intrauterine Device (IUD), or barrier and spermicide). Abstinence only is not an acceptable method. Patients must agree to use adequate contraception during the study and for 4 weeks after their last dose of corticotrophin (ACTH). Male patients must agree to ensure they or their female partner(s) are using adequate contraception during the study and for 4 weeks after the patient receives their last dose of corticotrophin (ACTH).
4. Patients must have a new diagnosis of adult-onset rheumatoid arthritis (RA) as defined by the 2010 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria and who have had symptoms for <1 year.
5. Patients must be experiencing mild to moderate rheumatoid arthritis ( RA), have at least 6 tender and 6 swollen joints at screening and a clinical disease activity index (CDAI) score of > 6.0
6. A Baseline Magnetic Resonance Imaging ( MRI) must show the presence of osteitis or erosions in the hand or wrist.
7. Patients must be able and willing to comply with the requirements of the study protocol.
8. Patients must have a C-reactive Protein (CRP) or erythrocyte sedimentation rate (ESR) > upper limits of normal

Exclusion criteria:

1. Patients who have a diagnosis of any other inflammatory arthritis (e.g., psoriatic arthritis or ankylosing spondylitis).
2. Patients with exposure to any disease modifying antirheumatic drug (DMARD), Biologic, Non-biologic or experimental medication for the treatment of rheumatoid arthritis (RA).
3. Patients with a non-inflammatory type of arthritis (e.g. osteoarthritis or fibromyalgia) that in the Investigator's opinion is symptomatic enough to interfere with evaluation of the effect of study drug on the patient's primary diagnosis of rheumatoid arthritis (RA).
4. Patients with history of an infected joint prosthesis at any time with that prosthesis still in situ.
5. Patients have received prohibited medication:

   * non-steroidal anti-inflammatory drug (NSAIDs /COX-2 inhibitors) (any change in dose regimen in the 7 days prior to baseline)
   * Oral corticosteroids within 4 weeks of baseline
   * Intra-muscular, intra-venous, intra-articular (IM/IV/IA) corticosteroids/ Intra-articular (IA) Hyaluronic acid (any dose 28 days prior to baseline)
6. Female patients who are breast-feeding, pregnant, or plan to become pregnant during the trial or within twelve weeks following last dose of study drug.
7. Patients with a history of chronic infection due to fungal, parasitic or mycotic pathogens during the preceding year, recent serious or life-threatening infection within 6 months (including herpes zoster), or any current sign or symptom that may indicate an infection.
8. Patients with active Tuberculosis (TB) (or history of active TB), positive chest X-ray for TB, or positive (defined as induration of ≥ 5mm) purified protein derivative (PPD) skin test, positive QuantiFERON, or patients having close contact with an individual with active TB. Patients having a PPD skin test ≥ 5 mm or a positive QuantiFERON test can enter the study, provided that active TB is excluded and provided that they are adequately treated for latent TB (e.g., isonicotinic acid hydrazide [INH therapy] for 9 months [with vitamin B6]) and provided that appropriate treatment is initiated simultaneously with the first administration of ACTH.
9. Patients at a high risk of infection (e.g. leg ulcers, indwelling urinary catheter and persistent or recurrent chest infections and patients who are permanently bedridden or wheelchair bound).
10. Patients with a known allergy or intolerance to steroids 11 Concurrent malignancy or a history of malignancy (other than carcinoma of the cervix or basal cell carcinoma successfully treated more than 5 years prior to screening).

12. Patients with a current or recent history of severe, progressive, and/or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological or cerebral disease.

13. Patients with class III or IV congestive heart failure according to the New York Heart Association (NYHA) 1964 classification criteria.

14. Patients with a history of, or suspected, demyelinating disease of the central nervous system (e.g. multiple sclerosis or optic neuritis).

15. Patients with any other condition (e.g. clinically significant laboratory values) which in the Investigator's judgment would make the patient unsuitable for inclusion in the study.

16. Patients who have a metal device affected by MRI (e.g., any type of electronic, mechanical, or magnetic implant; cardiac pacemaker; aneurysm clip(s); implanted cardioverter defibrillator; or a cochlear implant) 17. Patients who have a potential ferromagnetic foreign body (metal slivers, metal shavings, other metal objects) for which they have sought medical attention.

18. Concurrent steroid use for any concomitant disease. 19. Subjects who are known to be Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman B Gaylis, MD, Principal Investigator — AARDS Research, Inc.
Locations (1):
- AARDS Research, Inc, Aventura, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Ten (10) Patients were treated with 80 U of ACTH once weekly and MTX 12.5-25 mg/week for a period of 6 months. Eight (8) Patients completed the 6 month trial in this group
- Group 2: Ten (10) patients were treated with 80 U of ACTH twice a week and MTX 12.5-25 mg/week for a 6 month period. Nine (9) patients completed the trial in this group over the 6 month period.
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 10 | 10
Completed | 8 | 9
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Corticotrophin 80 Units | Corticotrophin 80 Units Twice a Week | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Full Range); unit: years] | 60 [49 to 77] | 57 [36 to 78] | 59 [36 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Score
Description: To evaluate the effect of the use of 2 doses of corticotrophin (ACTH) as a treatment in patients with early onset rheumatoid arthritis as an alternative to conventional steroid therapy by evaluating the change from baseline in the clinical findings as measured by Clinical Disease Activity Index (CDAI) scores. The CDAI is calculated at the specified time points using the formula: CDAI = SJC(28) + TJC(28) + PGA + EGA SJC(28): Swollen 28-Joint Count (shoulders, elbows, wrists, MCPs, PIPs including thumb IP, knees) Interpretation: A lower CDAI score from Baseline would mean improvement in disease activity and an increase in CDAI score from Baseline would mean an increase in disease activity or a worsening in disease activity. Scores: 0.0-2.8 = Range for Remission; 2.9-10.0 = Range for Low disease activity; 10.1-22.0 Range for Moderate disease activity; 22.1-76 Range for High disease activity.Total range is from 0-100, with the high scores representing high disease activity.
Time Frame: Baseline, Month 3 and Month 6
Population: Total number of Patients who complete 6 months of treatment in both groups doses weekly Group 1, and dosed twice a week Group 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 9 | 8
Participants
  Baseline: remission | 0 | 0
  Baseline: low disease activity | 0 | 0
  Baseline: moderate disease activity | 0 | 0
  Baseline: high disease activity | 9 | 8
  Month 3: remission | 3 | 1
  Month 3: low disease activity | 2 | 4
  Month 3: moderate disease activity | 4 | 2
  Month 3: high disease activity | 0 | 1
  Month 6: remission | 2 | 3
  Month 6: low disease activity | 4 | 3
  Month 6: moderate disease activity | 2 | 2
  Month 6: high disease activity | 1 | 0

2. Secondary Outcome: Evaluation of MRI Structural Improvements
Description: To compare the number of patients who have synovitis, oseitis and erosions at Baseline, Month 3 and Month 6. Normal range for synovitis, osteitis and erosions is zero (0)
Time Frame: Baseline, 3 months, 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Group 1: Patients being weekly dosed with ACTH at 80 units
- Group 2: Patients receiving twice weekly doing of 80 units ACTH
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 9 | 8
participants
  Baseline : synovitis | 8 | 7
  Baseline : osteitis | 8 | 4
  Baseline : erosions | 9 | 8
  Month 3 : synovitis | 6 | 7
  Month 3 : osteitis | 6 | 6
  Month 3 : erosions | 9 | 8
  Month 6 : synovitis | 5 | 7
  Month 6 : osteitis | 4 | 4
  Month 6 : erosions | 7 | 8

3. Secondary Outcome: Number of Participants With Increased or Decreased Erosions of the Hand and Wrist
Description: Comparison of the change in the number of erosions seen in the joints of the hand and wrist as measured by Magnetic Resonance Imaging (MRI) findings.
  Regression indicates improvement in the number of erosions seen from Baseline and Progression indicates worsening in the number of erosions seen from Baseline. Normal range is zero (0).
Time Frame: Month 3 and Month 6
Population: Total number of Patients with erosions who completed 6 months of treatment in both groups doses weekly Group 1, and dosed twice a week Group 2
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 9 | 8
participants
  Month 3 : Progressed erosions | 1 | 3
  Month 3 : Regressed erosions | 0 | 2
  Month 6 : Progressed erosions | 2 | 2
  Month 6 : Regressed erosions | 1 | 2

4. Secondary Outcome: Comparison of Clinical Disease Activity Index (CDAI) Scores to Positive Magnetic Resonance Imaging (MRI) Findings
Description: Comparison of the clinical findings as measured by the Clinical Disease Activity Index (CDAI) versus the structural findings as measured by Magnetic Resonance Imaging (MRI). Improvement is measured as a reduction in CDAI score from Baseline to Month 6 and improvement in MRI is regression of erosions, oseitis and synovitis at month 6. Norman MRI score is zero (0).
  CDAI: 0.0-2.8 remission; 2.9-10.0 low disease activity; 10.1-22 moderate disease activity; 22.1-76 high disease activity. A decrease in CDAI score is improvement
Time Frame: Month 6
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 9 | 8
participants
  # of patients whose CDAI score improved | 8 | 8
  # of patients whose overall MRI improved | 6 | 5

5. Other Pre Specified Outcome: Participants With Increased and Decreased C-Reactive Protein (CRP) Values and Erythrocyte Sedimentation Rates (ESR)
Description: comparisons not statistical analysis will be made from Baseline and Month 6 of the C- reactive Protein (CRP) values and Erythrocyte Sedimentation Rate (ESR) to determine the number of patients whose test result improved or worsenedCRP value (normal range <1.0 mg/dl). ESR (normal range 0-28 mm/hr) . If the value is increased, the disease activity worsened. If the value is reduced the disease activity is improved.
Time Frame: Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 9 | 8
Participants
  CRP Values: # of patient with Decreased values | 8 | 7
  CRP Values: # of patients with Increased values | 1 | 1
  ESR Values: # of patient with Decreased values | 9 | 8
  ESR Values: # of patients with Increased values | 0 | 0

ADVERSE EVENTS:
Time Frame: all adverse events were collected from the date of signing Informed Consent and Discontinuation or Completion of the trial. There were no adverse events either serious or non-serious to be reported.
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No